CLINICAL TRIAL: NCT05243186
Title: Assessing Cognitive Performance Among Adults With Attention Disorders Working on Treadmill
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ariel University (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ArielUni
Record Dates: First submitted 2022-01-23; First posted 2022-02-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-10

CONDITIONS: Attention Deficit Disorder
Keywords: Attention Deficit Disorder; Cognitive performance; Treadmill
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: All participants will participate in four different sessions of the study that will be randomly crossed over.
Masking Description: There are no masking in the study. All parties have all the information regard the conditions of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MPH walking (Experimental): The participants will be instructed to work while taking Methylphenidate and walking on a treadmill workstation
  Interventions: Device: Treadmill workstation; Drug: Methylphenidate
- MPH sitting (Placebo Comparator): The participants will be instructed to work while taking Methylphenidate and sitting at a desk
  Interventions: Drug: Methylphenidate
- No MPH walking (Placebo Comparator): The participants will be instructed to work without taking Methylphenidate while walking on a treadmill workstation
  Interventions: Device: Treadmill workstation
- No MPH sitting (Placebo Comparator): The participants will be instructed to work without taking Methylphenidate while sitting at a desk
  Interventions: Device: Treadmill workstation; Drug: Methylphenidate

INTERVENTIONS:
Device: Treadmill workstation — walking on a treadmill workstation next to desk with computer and screen
  Other Names: Walking on a treadmill workstation
  Arms: MPH walking; No MPH sitting; No MPH walking
Drug: Methylphenidate — Using prescription drug
  Other Names: Ritalin
  Arms: MPH sitting; MPH walking; No MPH sitting

SUMMARY:
Randomized clinical trial in which individuals who have been diagnosed with ADHD and are regularly treated with Methylphenidate will be test for cognitive performance and will be randomly examined in the following four conditions:

* While taking Methylphenidate and sitting at a desk
* While taking Methylphenidate and walking on a treadmill workstation
* Without taking Methylphenidate while sitting at a desk
* Without taking Methylphenidate while walking on a treadmill workstation The investigators will compare the cognitive achievements outcomes and evaluate the efficiency of studying in each of these four conditions.

DETAILED DESCRIPTION:
The rationale of this clinical trial is to identify the intervention that best contributes to better cognition results of adults with ADHD's: physical activity, drug or a combination of the two? The study will enable to determine which factor will improve cognitive results. The findings of this trial will help determine the best treatment method that can be offer to adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Insured by Maccabi Health Services

* Diagnosed with ADHD by Neurologist/Psychiatrist/Developmental Doctor
* Take Methylphenidate as part of the treatment for ADHD AND have agreed to not take the drug if asked to
* Understand the language and simple instruction
* Willing to participate in the study and sign the agreement form

Exclusion Criteria:

* Suffer from heart disease or chronic respiratory illness
* Women who are pregnant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Stroop performance | Through study completion, an average of 1 year
  The Stroop task measures selectivity and distraction and evaluate the inhibitory ability. In this task a word is displayed in two coloured rectangles. Three states are included: Neutral state- where the word is colored in black; Congruent state- word's meaning and its color correspond; Non-congruent state- word's meaning does not match the color. For each state, parameters are shown separately. Calculated parameters include Mean reaction time of correct responses± the standard deviation of correct reaction times and errors- number of incorrect responses, where subjects pressed the wrong key. The scale of mean response time displays the mean score number of milliseconds for a subject to response (higher number present longer time of response- worse outcome). Higher standard deviation indicates larger distribution among the averages of the subjects. Errors count the times that subjects made mistakes in their answers starting from zero- higher score means worse outcome.
Barhatt performance | Through study completion, an average of 1 year
  Barhatt performance is a validated questionnaire that includ 30 statements designed to assess impulsivity. The values on a 4-point scale rang from 1 ("never/rarely "), 2 ("sometimes"), 3 ("frequently"), and 4 ("almost always/always"). These statements create three subscales/ dimensions: 1. Motor Impulsiveness (MI), which reflects action without forethought (for example, "I do things without thinking"), 2. Attentional Impulsiveness (AI), which reflects a reduced ability to maintain attention toward a stimulus (for example, "I concentrate easily"), and 3. Non-Planning Impulsiveness (N-PI), which reflects an emphasis on the present (for example, "I am more interested in the present than the future"). In all these three dimensions higher mean score represent higher impulsivity.
Breaks from work | Through study completion, an average of 1 year
  Number and length of breaks the participants took from their cognitive work. The values represent the mean number of breaks subjects took during their working time, higher numbers represent more breaks. As well the mean time of breaks in minutes where higher number represents longer time of break.

CONTACTS AND LOCATIONS:
Overall Officials: Liat Korn, PhD, Principal Investigator — Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Yes
The result of the study will be analyzed. A paper will be submitted to an international journal with study description including methods, examination protocol results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year
Access Criteria: Pending collaborators decision.

REFERENCES:
- [Background] Korn L, Hassan K, Fainshtein N, Yusov N, Davidovitch N. Non-Medical Use of Prescription Stimulants for Treatment of Attention Disorders by University Students: Characteristics and Associations. Med Sci Monit. 2019 May 21;25:3778-3787. doi: 10.12659/MSM.913973. PMID 31111829